CLINICAL TRIAL: NCT03696797
Title: Iron Reduction by Phlebotomy for the Treatment of Diabetes and Nonalcoholic Fatty Liver Disease
Brief Title: Iron Reduction for the Treatment of Diabetes and Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00044393; 1R01DK119913-01 (NIH)
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-07

CONDITIONS: Iron; Diabetes; Nonalcoholic Fatty Liver
Keywords: Iron Reduction; Phlebotomy
MeSH Terms: conditions — Diabetes Mellitus; Non-alcoholic Fatty Liver Disease | interventions — Blood Donation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Both groups will not know assignment as all will have a sleep mask (like a blindfold, covering the eyes, held on with an elastic band) placed so participant will not know whether blood was actually removed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): Will have a Unit of blood (two cups, the same amount donated at the Red Cross) drawn. This involves having a needle inserted into a vein in your arm. Prior to taking the blood, staff will measure your blood count to be sure you are not anemic, and blood pressure to be sure no dehydration. During or after donation, a sports drink is provided to replace the fluid loss. Phlebotomy
  Interventions: Procedure: Blood Donation
- Control Group (Sham Comparator): Will not donate blood, but will have a needle inserted into a vein in your arm. Both groups will not know which group assignment they have been randomized. Sham Phlebotomy
  Interventions: Procedure: Sham Blood Donation

INTERVENTIONS:
Procedure: Blood Donation — Participants in the TREATMENT GROUP will have a Unit of blood (two cups, the same amount you would donate at the Red Cross) drawn. This involves having a needle inserted into a vein in your arm. Prior to taking the blood, staff will measure blood count to be sure participants are not anemic, and blood pressure to be sure there is no dehydration. During or after donation, participants will be given a sports drink to replace the fluid loss. Participants in the CONTROL GROUP will not donate blood, but will have a needle inserted into a vein in your arm. Neither group will not know to which they have been assigned, all will have a sleep mask (like a blindfold, covering the eyes, held on with an elastic band) placed so they will not know whether blood was actually removed.
  Arms: Treatment Group
Procedure: Sham Blood Donation — Participants will have a needle inserted their arm, however, no blood will be drawn.
  Arms: Control Group

SUMMARY:
This is a treatment study to determine if reducing the body's iron stores by blood donation will improve diabetes control and other problems associated with diabetes such as fatty liver disease.

DETAILED DESCRIPTION:
Investigators propose that high iron triggers a number of events in different tissues, some of which will predispose to diabetes. Investigators will therefore study normal individuals who have higher than average iron levels in tissues, test your glucose control through standard blood tests like the hemoglobin A1c and by placing a continuous glucose monitor before and after participants have donated blood to determine if decreasing iron levels had any effect.

In addition, iron may also play a role in the progression of fatty liver to scarring and cirrhosis. Since 75% of people with diabetes have some degree of fatty liver, investigators would also like to study how the liver reacts to the lowering of iron.

There will be two optional sub studies conducted only at Wake Forest University Health Sciences they are: 1) Liver substudy that will look at liver complication of diabetes and the role it plays in the progression of fatty liver to scarring and cirrhosis. Investigators will look at how liver reacts to the lowering of iron. 2)Glucose Tolerance Mechanism substudy that will look at the mechanism the body uses to regulate blood sugar levels by insulin, this will require the frequently sample intravenous glucose tolerance test (FSIVGTT).

ELIGIBILITY:
Inclusion Criteria:

* Ages 40-75
* At least 3 months since diagnosis of prediabetes or diabetes
* HgbA1C value within three months or at screening of 5.7-6.4% for those with prediabetes and 7- 8.5% for those with diabetes (the upper limit of the latter to reduce the likelihood of major changes in glycemic intervention during the trial period, and the lower limit to allow some room for improvement)
* Undiagnosed on no medication HgA1C 6.5-6.9
* C-reactive protein levels up to 11.0
* Aim 2-serum ALT> 1.5 times the upper limit of normal, or; liver stiffness of > 12.5 kPa by Fibroscan transient elastography
* Serum ferritin levels within 1 year or at the time of screening in the upper half of the normal range (>50 ng/mL for women; >100ng/mL for men)

Exclusion Criteria:

* Documented anemia
* Hemoglobin levels within 0.5 g/dL of the lower limit of normal (<12.5 g/dL for women; 13.5 g/dL for men)
* Recent blood loss
* Bleeding diatheses (coagulation abnormalities or treatment with anticoagulants)
* Serious chronic infections or chronic inflammatory conditions that could elevate ferritin as an "acute phase reactant
* C-reactive protein greater than the upper limit of normal to further validate the lack of significant chronic inflammation
* Active cancer diagnosis (excluding skin cell cancers other than melanoma)
* Renal insufficiency (eGFR<60 ml/min)
* History of orthostatic hypotension
* Heavy alcohol use (NIH criteria for men, greater than 4 drinks on any day or 14/week)
* Pregnancy or premenopausal women of childbearing age, unless unable to become pregnant because of oral contraceptive use or surgical loss of ovaries or uterus
* Aim 2 - individuals meeting the additional inclusion criteria for aim 2 will be tested for anti-HAV IgM, HBs Ag, anti-HBc. IgM, anti HCV IgM and IgG. Subjects who prove positive for any of these viral serologies, except for HCV IgG will be excluded. The latter will be tested for HCV RNA by PRC, and if negative they will be eligible for enrollment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Change in HgbA1C | Baseline, Month 6
  Change in glycemia as measured byHgbA1C. Values from baseline and month 6 will be reported.
Change in ALT | Baseline, Month 12
  ALT values from baseline and month 12 will be reported.
Change in FSIGTT DI (Frequently sampled intravenous glucose tolerance test) | Baseline, Month 6
  FSIGTT DI Values from baseline and month 6 will be reported.

SECONDARY OUTCOMES:
HgbA1C at Month 12 | Month 12
  HgbA1C values will be reported.
Change in fasting glucose | Month 6, Month 12
  Fasting glucose measured on glucose machine (Abbott Freestyle Libre Pro system). Values of month 6 and month 12 will be reported.
Change in HOMA-IR (Homeostatic Model Assessment-Insulin Resistance) | Baseline, 12 months
  Insulin sensitivity measured by HOMA-IR (Homeostatic Model Assessment-Insulin Resistance) calculated from fasting glucose and insulin. Values will be reported for Baseline and 12 months.
Number of participants that Discontinued of oral antihyperglycemic agent | Month 12
  The numbers of participants that discontinued of oral antihyperglycemic agents
Change in Weight | Baseline, Month 12
  The change in weight from baseline to month 12 will be reported
Change in Blood Pressure | Baseline, Month 12
  The change in Blood pressure from baseline to month 12 will be reported
Number of participants that converted from pre-diabetes to Diabetes | Month 12
  Number of participants that converted from pre-Diabetes to Diabetes based on the HbA1C criteria.
Number of participants that converted from pre-diabetes to normal glucose tolerance | Month 12
  Number of participants that converted from pre-Diabetes to normal glucose tolerance based on the HbA1C criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Donald A McClain, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill (UNC), Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buysschaert M, Paris I, Selvais P, Hermans MP. Clinical aspects of diabetes secondary to idiopathic haemochromatosis in French-speaking Belgium. Diabetes Metab. 1997 Sep;23(4):308-13. PMID 9342544
- [Background] Abraham D, Rogers J, Gault P, Kushner JP, McClain DA. Increased insulin secretory capacity but decreased insulin sensitivity after correction of iron overload by phlebotomy in hereditary haemochromatosis. Diabetologia. 2006 Nov;49(11):2546-51. doi: 10.1007/s00125-006-0445-7. Epub 2006 Sep 22. PMID 17019598
- [Background] Bulaj ZJ, Ajioka RS, Phillips JD, LaSalle BA, Jorde LB, Griffen LM, Edwards CQ, Kushner JP. Disease-related conditions in relatives of patients with hemochromatosis. N Engl J Med. 2000 Nov 23;343(21):1529-35. doi: 10.1056/NEJM200011233432104. PMID 11087882
- [Background] Dmochowski K, Finegood DT, Francombe W, Tyler B, Zinman B. Factors determining glucose tolerance in patients with thalassemia major. J Clin Endocrinol Metab. 1993 Aug;77(2):478-83. doi: 10.1210/jcem.77.2.8345055.
- [Background] Ford ES, Cogswell ME. Diabetes and serum ferritin concentration among U.S. adults. Diabetes Care. 1999 Dec;22(12):1978-83. doi: 10.2337/diacare.22.12.1978. PMID 10587829
- [Background] Jiang R, Manson JE, Meigs JB, Ma J, Rifai N, Hu FB. Body iron stores in relation to risk of type 2 diabetes in apparently healthy women. JAMA. 2004 Feb 11;291(6):711-7. doi: 10.1001/jama.291.6.711. PMID 14871914
- [Background] Fleming DJ, Tucker KL, Jacques PF, Dallal GE, Wilson PW, Wood RJ. Dietary factors associated with the risk of high iron stores in the elderly Framingham Heart Study cohort. Am J Clin Nutr. 2002 Dec;76(6):1375-84. doi: 10.1093/ajcn/76.6.1375. PMID 12450906
- [Background] Afkhami-Ardekani M, Rashidi M. Iron status in women with and without gestational diabetes mellitus. J Diabetes Complications. 2009 May-Jun;23(3):194-8. doi: 10.1016/j.jdiacomp.2007.11.006. Epub 2008 Apr 16. PMID 18413178
- [Background] Wilson JG, Lindquist JH, Grambow SC, Crook ED, Maher JF. Potential role of increased iron stores in diabetes. Am J Med Sci. 2003 Jun;325(6):332-9. doi: 10.1097/00000441-200306000-00004. PMID 12811229
- [Background] Qiu C, Zhang C, Gelaye B, Enquobahrie DA, Frederick IO, Williams MA. Gestational diabetes mellitus in relation to maternal dietary heme iron and nonheme iron intake. Diabetes Care. 2011 Jul;34(7):1564-9. doi: 10.2337/dc11-0135. PMID 21709295
- [Background] Bowers K, Yeung E, Williams MA, Qi L, Tobias DK, Hu FB, Zhang C. A prospective study of prepregnancy dietary iron intake and risk for gestational diabetes mellitus. Diabetes Care. 2011 Jul;34(7):1557-63. doi: 10.2337/dc11-0134. PMID 21709294
- [Background] Sharifi F, Nasab NM, Zadeh HJ. Elevated serum ferritin concentrations in prediabetic subjects. Diab Vasc Dis Res. 2008 Mar;5(1):15-8. doi: 10.3132/dvdr.2008.003. PMID 18398807
- [Background] Jehn M, Clark JM, Guallar E. Serum ferritin and risk of the metabolic syndrome in U.S. adults. Diabetes Care. 2004 Oct;27(10):2422-8. doi: 10.2337/diacare.27.10.2422. PMID 15451911
- [Background] Fargion S, Mattioli M, Fracanzani AL, Sampietro M, Tavazzi D, Fociani P, Taioli E, Valenti L, Fiorelli G. Hyperferritinemia, iron overload, and multiple metabolic alterations identify patients at risk for nonalcoholic steatohepatitis. Am J Gastroenterol. 2001 Aug;96(8):2448-55. doi: 10.1111/j.1572-0241.2001.04052.x. PMID 11513189
- [Background] Altamura S, Muckenthaler MU. Iron toxicity in diseases of aging: Alzheimer's disease, Parkinson's disease and atherosclerosis. J Alzheimers Dis. 2009;16(4):879-95. doi: 10.3233/JAD-2009-1010. PMID 19387120
- [Background] Toyokuni S. Role of iron in carcinogenesis: cancer as a ferrotoxic disease. Cancer Sci. 2009 Jan;100(1):9-16. doi: 10.1111/j.1349-7006.2008.01001.x. Epub 2008 Oct 23. PMID 19018762
- [Background] Zhang W, Iso H, Ohira T, Date OC, Tanabe N, Kikuchi S, Tamakoshi A. Associations of dietary iron intake with mortality from cardiovascular disease: the JACC study. J Epidemiol. 2012;22(6):484-93. doi: 10.2188/jea.je20120006. Epub 2012 Sep 15. PMID 22986645
- [Background] Forouhi NG, Harding AH, Allison M, Sandhu MS, Welch A, Luben R, Bingham S, Khaw KT, Wareham NJ. Elevated serum ferritin levels predict new-onset type 2 diabetes: results from the EPIC-Norfolk prospective study. Diabetologia. 2007 May;50(5):949-56. doi: 10.1007/s00125-007-0604-5. Epub 2007 Mar 2. PMID 17333112
- [Background] Fargnoli JL, Fung TT, Olenczuk DM, Chamberland JP, Hu FB, Mantzoros CS. Adherence to healthy eating patterns is associated with higher circulating total and high-molecular-weight adiponectin and lower resistin concentrations in women from the Nurses' Health Study. Am J Clin Nutr. 2008 Nov;88(5):1213-24. doi: 10.3945/ajcn.2008.26480. PMID 18996855
- [Background] Gabrielsen JS, Gao Y, Simcox JA, Huang J, Thorup D, Jones D, Cooksey RC, Gabrielsen D, Adams TD, Hunt SC, Hopkins PN, Cefalu WT, McClain DA. Adipocyte iron regulates adiponectin and insulin sensitivity. J Clin Invest. 2012 Oct;122(10):3529-40. doi: 10.1172/JCI44421. Epub 2012 Sep 10. PMID 22996660
- [Background] Cooksey RC, Jones D, Gabrielsen S, Huang J, Simcox JA, Luo B, Soesanto Y, Rienhoff H, Abel ED, McClain DA. Dietary iron restriction or iron chelation protects from diabetes and loss of beta-cell function in the obese (ob/ob lep-/-) mouse. Am J Physiol Endocrinol Metab. 2010 Jun;298(6):E1236-43. doi: 10.1152/ajpendo.00022.2010. Epub 2010 Mar 30. PMID 20354157
- [Background] Houschyar KS, Ludtke R, Dobos GJ, Kalus U, Broecker-Preuss M, Rampp T, Brinkhaus B, Michalsen A. Effects of phlebotomy-induced reduction of body iron stores on metabolic syndrome: results from a randomized clinical trial. BMC Med. 2012 May 30;10:54. doi: 10.1186/1741-7015-10-54. PMID 22647517
- [Background] Fernandez-Real JM, Penarroja G, Castro A, Garcia-Bragado F, Hernandez-Aguado I, Ricart W. Blood letting in high-ferritin type 2 diabetes: effects on insulin sensitivity and beta-cell function. Diabetes. 2002 Apr;51(4):1000-4. doi: 10.2337/diabetes.51.4.1000. PMID 11916918
- [Background] Gao Y, Li Z, Gabrielsen JS, Simcox JA, Lee SH, Jones D, Cooksey B, Stoddard G, Cefalu WT, McClain DA. Adipocyte iron regulates leptin and food intake. J Clin Invest. 2015 Sep;125(9):3681-91. doi: 10.1172/JCI81860. Epub 2015 Aug 24. PMID 26301810
- [Background] Kusminski CM, Holland WL, Sun K, Park J, Spurgin SB, Lin Y, Askew GR, Simcox JA, McClain DA, Li C, Scherer PE. MitoNEET-driven alterations in adipocyte mitochondrial activity reveal a crucial adaptive process that preserves insulin sensitivity in obesity. Nat Med. 2012 Oct;18(10):1539-49. doi: 10.1038/nm.2899. Epub 2012 Sep 9. PMID 22961109
- [Background] Kowdley KV, Belt P, Wilson LA, Yeh MM, Neuschwander-Tetri BA, Chalasani N, Sanyal AJ, Nelson JE; NASH Clinical Research Network. Serum ferritin is an independent predictor of histologic severity and advanced fibrosis in patients with nonalcoholic fatty liver disease. Hepatology. 2012 Jan;55(1):77-85. doi: 10.1002/hep.24706. Epub 2011 Dec 6. PMID 21953442
- [Background] Valenti L, Fracanzani AL, Bugianesi E, Dongiovanni P, Galmozzi E, Vanni E, Canavesi E, Lattuada E, Roviaro G, Marchesini G, Fargion S. HFE genotype, parenchymal iron accumulation, and liver fibrosis in patients with nonalcoholic fatty liver disease. Gastroenterology. 2010 Mar;138(3):905-12. doi: 10.1053/j.gastro.2009.11.013. Epub 2009 Nov 18. PMID 19931264
- [Background] Duvnjak M, Barsic N, Tomasic V, Lerotic I. Genetic polymorphisms in non-alcoholic fatty liver disease: clues to pathogenesis and disease progression. World J Gastroenterol. 2009 Dec 28;15(48):6023-7. doi: 10.3748/wjg.15.6023. PMID 20027673
- [Background] Beaton MD, Chakrabarti S, Adams PC. Inflammation is not the cause of an elevated serum ferritin in non-alcoholic fatty liver disease. Ann Hepatol. 2014 May-Jun;13(3):353-6. PMID 24756010
- [Background] Valenti L, Fracanzani AL, Dongiovanni P, Rovida S, Rametta R, Fatta E, Pulixi EA, Maggioni M, Fargion S. A randomized trial of iron depletion in patients with nonalcoholic fatty liver disease and hyperferritinemia. World J Gastroenterol. 2014 Mar 21;20(11):3002-10. doi: 10.3748/wjg.v20.i11.3002. PMID 24659891
- [Background] Dongiovanni P, Fracanzani AL, Fargion S, Valenti L. Iron in fatty liver and in the metabolic syndrome: a promising therapeutic target. J Hepatol. 2011 Oct;55(4):920-32. doi: 10.1016/j.jhep.2011.05.008. Epub 2011 Jun 28. PMID 21718726
- [Background] Murali AR, Gupta A, Brown K. Systematic review and meta-analysis to determine the impact of iron depletion in dysmetabolic iron overload syndrome and non-alcoholic fatty liver disease. Hepatol Res. 2018 Feb;48(3):E30-E41. doi: 10.1111/hepr.12921. Epub 2017 Jul 20. PMID 28593739
- [Background] Adams LA, Crawford DH, Stuart K, House MJ, St Pierre TG, Webb M, Ching HL, Kava J, Bynevelt M, MacQuillan GC, Garas G, Ayonrinde OT, Mori TA, Croft KD, Niu X, Jeffrey GP, Olynyk JK. The impact of phlebotomy in nonalcoholic fatty liver disease: A prospective, randomized, controlled trial. Hepatology. 2015 May;61(5):1555-64. doi: 10.1002/hep.27662. Epub 2015 Mar 20. PMID 25524401
- [Background] Lorenzo C, Wagenknecht LE, Rewers MJ, Karter AJ, Bergman RN, Hanley AJ, Haffner SM. Disposition index, glucose effectiveness, and conversion to type 2 diabetes: the Insulin Resistance Atherosclerosis Study (IRAS). Diabetes Care. 2010 Sep;33(9):2098-103. doi: 10.2337/dc10-0165. PMID 20805282
- [Background] Koziol JA, Ho NJ, Felitti VJ, Beutler E. Reference centiles for serum ferritin and percentage of transferrin saturation, with application to mutations of the HFE gene. Clin Chem. 2001 Oct;47(10):1804-10. PMID 11568090
- [Background] Cheng HL, Bryant C, Cook R, O'Connor H, Rooney K, Steinbeck K. The relationship between obesity and hypoferraemia in adults: a systematic review. Obes Rev. 2012 Feb;13(2):150-61. doi: 10.1111/j.1467-789X.2011.00938.x. Epub 2011 Oct 10. PMID 21981048
- [Background] Ausk KJ, Ioannou GN. Is obesity associated with anemia of chronic disease? A population-based study. Obesity (Silver Spring). 2008 Oct;16(10):2356-61. doi: 10.1038/oby.2008.353. Epub 2008 Jul 24. PMID 18719644
- [Background] Andrews Guzman M, Arredondo Olguin M. Association between ferritin, high sensitivity C-reactive protein (hsCRP) and relative abundance of Hepcidin mRNA with the risk of type 2 diabetes in obese subjects. Nutr Hosp. 2014 Sep 1;30(3):577-84. doi: 10.3305/nh.2014.30.3.7647. PMID 25238834
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Beutler E, Felitti V, Ho NJ, Gelbart T. Relationship of body iron stores to levels of serum ferritin, serum iron, unsaturated iron binding capacity and transferrin saturation in patients with iron storage disease. Acta Haematol. 2002;107(3):145-9. doi: 10.1159/000057632. PMID 11978935

DOCUMENTS (1):
  • Informed Consent Form (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT03696797/ICF_000.pdf